CLINICAL TRIAL: NCT00521755
Title: Evaluation of Safety and Efficacy of Using Seraffix LTB - (Laser Tissue Bonding) System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seraffix (Industry)
Responsible Party: Dr. Hanna Levy, Clinical Study Consultant, Seraffix
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SF-01
Record Dates: First submitted 2007-08-26; First posted 2007-08-28 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2009-06

CONDITIONS: Dehiscence, Surgical Wound
Keywords: Laser bonding soft tissue albumin
MeSH Terms: conditions — Surgical Wound Dehiscence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Device: Seraffix LTB

INTERVENTIONS:
Device: Seraffix LTB — laser soldering for soft tissue wounds

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of using Seraffix LTB system for soft tissue bonding.

DETAILED DESCRIPTION:
Dermatologic wounds can be closed by a variety of methods. The choice of a particular closure technique should be based on the patient, wound, tissue characteristics, and anatomic location. The purpose of these closure methods is an approximation of wound lips until the regenerate tissue reach a phase, where it is closed and can sustain the daily tensile forces.

Several methods are used for wounds closure such as sutures, staples, tapes, tissue adhesives and laser energy. There have been two fundamental approaches to laser assisted bonding of tissues:

1. Laser welding-heating the approximated edges of cuts in tissues by a laser beam;
2. Laser soldering- applying a biological solder onto the approximated edges and heating the solder (and the underlying tissue).

Seraffix has developed the Seraffix LTB (Laser Tissue Bonding) System - a laser system for soft tissue bonding. This innovative system includes features that make laser soldering suitable for clinical use. The Seraffix system is composed of CO2 laser device, propriety grip device (Clamps) and soldering agent (Human Albumin).

ELIGIBILITY:
Inclusion Criteria:

* Male/Female age 18-60.
* Subject is scheduled for laparoscopic cholecystectomy surgery.
* Subject able to comprehend and give informed consent for participation in this study.
* Signed informed consent form.

Exclusion Criteria:

* Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months prior to screening.
* Acute infection requiring intravenous antibiotics at the time of screening.
* Bleeding, coagulation and or clotting disorders.
* Diabetes mellitus: IDDM or NIDDM.
* HIV positive or any other immunosuppressive disorder.
* Renal failure (Serum creatinine >2.0 mg/dl).
* Inflammatory and or allergic diseases or condition of the skin: Psoriasis, Eczema or dermatitis.
* Any concomitant infection - viral or bacterial.
* Drug abuse.
* Use of steroids.
* Infection / abscess / pain in treatment target area.
* Pregnancy or lactating.
* History of keloid scarring.
* Use of aspirin or antioxidants
* Subject is suffering extreme general weakness.
* Subject objects to the study protocol.
* Known cognitive or psychiatric disorder
* Concurrent participation in any other clinical study.
* Physician objection.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-11 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Primary study endpoint will be to establish the safety of using the Seraffix System for tissue bonding and wounds closure. Safety will be established by paucity of serious adverse events and adverse events. | 3 months

SECONDARY OUTCOMES:
1. Re-intervention: A subject is scored a success (1) if he had No Re-intervention by 3 months; otherwise he is scored a failure (0). 2. Wound dehiscence of at least 50% of wound length: | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ossama Hatoum, Dr., Principal Investigator — HaEmek Medical Center, Israel
Locations (1):
- Haemek Medical Center, Afula, Israel